CLINICAL TRIAL: NCT04640649
Title: A Novel Approach to Personalized Prediction of Progression of Age-Related Macular Degeneration
Brief Title: Prediction of Progression of Age-Related Macular Degeneration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Stanford University (Other); Illinois Retina Associates (Other); Bascom Palmer Eye Institute (Other)
Responsible Party: Principal Investigator, Joelle Hallak, Assistant Professor, Director, University of Illinois at Chicago
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-0460
Record Dates: First submitted 2020-10-08; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Macular Degeneration; Macular Degeneration, Wet; Macular Degeneration, Dry
MeSH Terms: conditions — Macular Degeneration; Wet Macular Degeneration; Geographic Atrophy | interventions — Prediction Algorithms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prediction Algorithm (Experimental): Patients in the test arm will have a screening visit, then will come for two follow-up visits, at 3 months (if the algorithm determines high-risk of conversion within 3 months) and 6 months.
  Interventions: Other: Algorithm prediction
- Control (No Intervention): Patients in the control arm will have a screening visit, then will come for one follow-up visit, at 6 months (standard care) only.

INTERVENTIONS:
Other: Algorithm prediction — Patients with early and intermediate AMD in at least one eye who are at risk of converting to wet AMD or GA expansion will be randomly assigned to a test group or control group. The test group will have their baseline data analyzed by an algorithm to predict the probability of conversion to wet AMD. If the probability is high for conversion at or before 3 months, patients will have earlier follow-up care than the control group (standard follow-up care every 6 months).
  Arms: Prediction Algorithm

SUMMARY:
The goal for this study is to initiate a randomized, controlled clinical trial to test the viability of personalized AMD progression prediction models. Early and intermediate AMD patients will be recruited and randomly assigned them to a control or test group. The test group will include patients who will receive personalized follow-up care based on their predicted risk, and collect baseline and follow-up data.

This work will advance the AMD field by improving the identification of high-risk patients as candidates for more frequent screening and earlier treatment, leading to better clinical outcomes.

DETAILED DESCRIPTION:
More than 90% of patients with advanced AMD have severe vision loss. Predicting AMD progression from an early or intermediate stage is crucial, since prompt intervention after a choroidal neovascularization (CNV) event and geographic atrophy (GA) monitoring can greatly improve visual outcomes. Patients at higher risk of progression should have more frequent follow-up visits, since progression often occurs before any visual changes are noticed by the patient. Previous work has determined the risk factors for AMD progression based on drusen features in fundus photos, Optical Coherence Tomography (OCT) and from genetic factors. However, current models are limited by their ability to make predictions over short intervals, which limits their utility in guiding screening intervals.

In this study we will recruit patients with early and intermediate AMD in at least one eye who are at risk of converting to wet AMD or GA expansion. We will perform a randomized trial where we will randomly assign them to a control or test group (personalized follow-up care starting at 3 months based on their predicted risk from algorithm results), and collect baseline genetic, demographic, imaging, and clinical data and first follow-up data at the 3 month and 6 month follow-up time points. Outcomes will be measured to determine if an algorithm predicting early follow-up for high-risk patients (3 month) is advantageous over the standard 6 month follow-up time point.

ELIGIBILITY:
Inclusion Criteria:

* Non-neovascular AMD at baseline in at least one eye with no signs of GA,
* > 45 years of age,
* willingness to participate through a signed consent form.

Exclusion Criteria:

* Pregnant women and vulnerable populations
* Participation in an investigational trial that involves treatment with any drug (with the exception of vitamins or minerals) within 3 months prior to Day 1.
* Any history of macular pathology unrelated to AMD affecting vision or contributing to the presence of intraretinal or subretinal fluid

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | one year
  The primary outcome measure will be the difference in visual acuity between test and control patients in those who progressed to late stage AMD

SECONDARY OUTCOMES:
Actual risk of conversion | one year
  The actual risk/ of conversion to wet AMD will be calculated for each eye that progressed using regression analysis. This risk will be compared to the risk that the algorithm predicted.
Number of visits | one year
  Number of visits will be compared between the test arm and the control arm of patients who progression to wet AMD

CONTACTS AND LOCATIONS:
Overall Officials: Joelle A Hallak, PhD, Principal Investigator — University of Illinois at Chicago

IPD SHARING:
Plan to Share IPD: No